CLINICAL TRIAL: NCT00426777
Title: A Randomized, Single-blind, Placebo-controlled, Multicentre Study to Evaluate the Effect of Risedronate and Placebo on Bone Mineral Density in Men Undergoing Androgen Deprivation Therapy With Leuprolide Acetate
Brief Title: Efficacy Study of Risedronate to Prevent Cancer Treatment-Induced Bone Loss in Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CMX Research (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SA-CMX-01
Record Dates: First submitted 2007-01-24; First posted 2007-01-25 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostatic adenoma; prostatic neoplasm
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- risedronate (Active Comparator)
  Interventions: Drug: risedronate
- placebo (Placebo Comparator)
  Interventions: Drug: Control

INTERVENTIONS:
Drug: risedronate — risedronate 35mg tablet, weekly for 12 months
  Other Names: Actonel
  Arms: risedronate
Drug: risedronate — 35mg weekly
  Other Names: Actonel
  Arms: risedronate
Drug: Control — risedronate-matched placebo weekly
  Arms: placebo

SUMMARY:
Prostate cancer patients treated with LHRH agonists (e.g., leuprolide) lose bone mineral density. This is similar to post-menopausal osteoporosis. Risedronate is approved to prevent osteoporosis. We hypothesize that risedronate may also be effective in prostate cancer patients treated with LHRH agonists.

DETAILED DESCRIPTION:
IV bisphosphonates have proven effective in treating bone loss in prostate cancer patients treated with LHRH agonists. However, it is yet to be determined if an oral bisphosphonate such as risedronate could offer the same benefits.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Histologically confirmed diagnosis of prostate cancer without metastases.
* Patient must have negative bone scan to rule out bone metastases.
* Patient for whom androgen deprivation therapy with leuprolide acetate is indicated for at least 1 year.
* Eastern Cooperative Oncology Group (ECOG) score of 0 - 2.
* Study medication must be started within 3 months of initiation of ADT.
* Signed written informed consent.

Exclusion Criteria:

* Prior ADT (greater than 3 months).
* History of treatment with calcitriol or bisphosphonates.
* Suppressive doses of thyroxine within the previous year.
* Concomitant or prior history of long-term treatment (greater than or equal to 3 months) with systemic glucocorticoids.
* Evidence of any of the following conditions per subject self-report or chart review:

Current hyper- or hypothyroidism (stable on thyroid replacement therapy is allowed, if TSH is within normal reference range).

Paget's disease, Cushing's disease, hyperprolactinemia, chronic liver disease. Unstable systemic disease including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months before randomization.

Major surgery or significant traumatic injury occurring within 1 month prior to randomization.

* Known hypersensitivity to leuprolide acetate or any of the components found in Eligard
* Any concurrent condition that would make it undesirable, in the physician's opinion, for the subject to participate in the study or would jeopardize compliance with the protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
bone mineral density of the lumbar spine | 12 months

SECONDARY OUTCOMES:
overall safety | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Casey, M.D., Principal Investigator — CMX Research
Locations (21):
- Canada (21):
  - Southern Interior Medical Research Corporation, Kelowna, British Columbia
  - Dr. Cal Andreou, Surrey, British Columbia
  - Dr. Allan Patrick, Fredericton, New Brunswick
  - The Male/Female Health and Research Centre, Barrie, Ontario
  - Dr. Stanley Flax, Brampton, Ontario
  - Brantford Urology Research, Medical Arts Building, Brantford, Ontario
  - G. Kenneth Jansz Medicine Professional Corporation, Burlington, Ontario
  - Urology Research Centre, Burlington, Ontario
  - Northern Urology Centre, Greater Sudbury, Ontario
  - Guelph Urology Associates, Guelph, Ontario
  - Credit Valley Medical Arts Centre, Mississauga, Ontario
  - Mor Urology Inc., Bayview Business Centre, Newmarket, Ontario
  - The Male and Female Health Centre, Oakville, Ontario
  - Orillia Urology Associates, Orillia, Ontario
  - Urotec, Oshawa, Ontario
  - Dr. Todd Webster, Owen Sound, Ontario
  - Kawartha Urology Associates, Peterborough, Ontario
  - Dr. Allan Abramovitch, Scarborough Village, Ontario
  - The Male Health Centre, Toronto, Ontario
  - Dr. Roger J. Buckley, Willowdale, Ontario
  - Urology South Shore Research, Greenfield Park, Quebec